CLINICAL TRIAL: NCT03155997
Title: A Randomized, Open-Label, Phase 3 Study of Abemaciclib Combined With Standard Adjuvant Endocrine Therapy Versus Standard Adjuvant Endocrine Therapy Alone in Patients With High Risk, Node Positive, Early Stage, Hormone Receptor Positive, Human Epidermal Receptor 2 Negative, Breast Cancer
Brief Title: Endocrine Therapy With or Without Abemaciclib (LY2835219) Following Surgery in Participants With Breast Cancer
Acronym: monarchE
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: NSABP Foundation Inc (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16338; I3Y-MC-JPCF (Other: Eli Lilly and Company); 2016-004362-26 (EudraCT Number); NSABP B-58 (Other: NSABP)
Expanded Access: NCT03763604 (Approved for marketing)
Record Dates: First submitted 2017-05-15; First posted 2017-05-16 (Actual); Results first posted 2021-04-09 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
Keywords: early stage breast cancer; cyclin-dependent kinase (CDK)
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 150 mg Abemaciclib + Endocrine Therapy (Experimental): Participants received Abemaciclib orally at 150 milligrams (mg) twice daily with at least 6 hours between doses for up to 2 years or until evidence of disease recurrence or other discontinuation criteria were met, whichever occurs first. Endocrine therapy (physicians' choice) standard-of-care was administered according to package label until discontinuation criteria were met.
  Interventions: Drug: Abemaciclib; Drug: Standard Adjuvant Endocrine Therapy
- Endocrine Therapy (Other): Endocrine therapy (physicians' choice) standard-of-care was administered according to package label until discontinuation criteria were met.
  Interventions: Drug: Standard Adjuvant Endocrine Therapy

INTERVENTIONS:
Drug: Abemaciclib — Administered orally.
  Other Names: LY2835219
  Arms: 150 mg Abemaciclib + Endocrine Therapy
Drug: Standard Adjuvant Endocrine Therapy — Administered according to label instructions.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the study drug abemaciclib in participants with high risk, node positive, early stage, hormone receptor positive (HR+), human epidermal receptor 2 negative (HER2-), breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women (regardless of menopausal status) or men ≥18 years of age (or per local regulations).
* The participant has confirmed HR+, HER2-, early stage resected invasive breast cancer without evidence of distant metastases.
* The participant must have undergone definitive surgery of the primary breast tumor.
* The participant must have tumor tissue from breast (preferred) or lymph node for exploratory biomarker analysis available prior to randomization.
* Pathologic lymph node involvement and at least one of the following indicating a higher risk of recurrence:

  * 4 or more positive axillary lymph nodes
  * Tumor size of at least 5 centimeters
  * Grade 3 defined as at least 8 points on the Bloom Richardson grading system
  * Ki-67 index by central analysis of ≥20% on untreated breast tissue
* The participant must be randomized within 16 months from the time of definitive breast cancer surgery.
* The participant may receive up to 12 weeks of endocrine therapy until randomization following the last non-endocrine therapy (surgery, chemotherapy, or radiation) whichever is last.
* Participants must have recovered (grade ≤1) from the acute effects of chemotherapy and radiotherapy and from surgical side effects following definitive breast surgery.
* Women of reproductive potential must have a negative blood pregnancy test and agree to use highly effective contraceptive methods.
* The participant has a Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
* The participant has adequate organ function.
* The participant is able to swallow oral medications.

Exclusion Criteria:

* Metastatic disease (including contralateral axillary lymph nodes) or node-negative disease.
* Participants with inflammatory breast cancer.
* Participants with a history of previous breast cancer, with the exception of ipsilateral ductal carcinoma in situ (DCIS) treated by locoregional therapy alone ≥5 years ago. Participants with a history of contralateral DCIS treated by local regional therapy at any time may be eligible. Participants with a history of any other cancer (except non-melanoma skin cancer or carcinoma in situ of the cervix), unless in complete remission with no therapy for a minimum of 5 years from the date of randomization are excluded.
* Females who are pregnant or lactating.
* The participant has previously received treatment with any CDK4 and CDK6 inhibitor.
* The participant is receiving concurrent exogenous reproductive hormone therapy (for example, birth control pills, hormone replacement therapy, or megestrol acetate).
* The participant has previously received endocrine therapy for breast cancer prevention (tamoxifen or aromatase inhibitors) or raloxifene.
* The participant has serious preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study.
* The participant has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin or sudden cardiac arrest. Any participant with a history of venous thromboembolism (VTE).
* The participant has active systemic infections or viral load.
* The participant has received an experimental treatment in a clinical trial within the last 30 days or 5 half-lives, whichever is longer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5637 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2029-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (619):
- United States (162):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Arizona Oncology Associates, P.C. - HOPE, Goodyear, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Mayo Clinic Hospital, Phoenix, Arizona
  - The University of Arizona Cancer Center, Tucson, Arizona
  - Yuma Regional Cancer Center, Yuma, Arizona
  - St. Bernards Medical Center, Jonesboro, Arkansas
  - Highlands Oncology Group, Springdale, Arkansas
  - Beverly Hills Cancer Center, Beverly Hills, California
  - Roy and Patricia Disney Family Cancer Center - Providence Saint Joseph Medical Center, Burbank, California
  - City of Hope National Medical Center, Duarte, California
  - California Cancer Associates Research and Excellence, Fresno, California
  - Kaiser Permanente, Harbor City, California
  - Loma Linda University School of Medicine, Loma Linda, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Pacific Cancer Care, Monterey, California
  - St. Joseph Hospital, Orange, California
  - University of California Davis (UC Davis) Comprehensive Cancer Center, Sacramento, California
  - UCSF Medical Center at Mission Bay, San Francisco, California
  - California Cancer Associates in Research and Excellence, San Marcos, California
  - Dignity Health Dominican Oncology and Hematology, Santa Cruz, California
  - Kaiser Permanente, Vallejo, California
  - USO-Rocky Mountain Cancer Center, Boulder, Colorado
  - USO-Rocky Mountain Cancer Center, Thornton, Colorado
  - Yale-New Haven Hospital, New Haven, Connecticut
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - University of Florida College of Medicine, Gainesville, Florida
  - Millennium Oncology - Hollywood, Hollywood, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Florida Cancer Specialists - North, Lecanto, Florida
  - Ocala Oncology, P.A., Ocala, Florida
  - Tallahassee Memorial Cancer Center, Tallahassee, Florida
  - Moffitt Cancer Center, Richard M. Shulze Family Foundation Outpatient Center, Tampa, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital, Marietta, Georgia
  - Summit Cancer Care DBA Candler Medical Oncology Practice, Savannah, Georgia
  - University of Hawaii Cancer Center, Honolulu, Hawaii
  - John H. Stroger Hospital of Cook County, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Edward Cancer Center, Naperville, Illinois
  - Quincy Medical Group, Quincy, Illinois
  - Franciscan St. Francis Health, Indianapolis, Indiana
  - Community Howard Oncology Center, Kokomo, Indiana
  - Cancer Center of Kansas, Wichita, Kansas
  - Univ of Louisville School of Medicine, Louisville, Kentucky
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - Terrebonne General Medical Center, Houma, Louisiana
  - Cancer Care of Maine, Brewer, Maine
  - New England Cancer Specialists - Kennebunk, Kennebunk, Maine
  - Central Maine Medical Center, Lewiston, Maine
  - Meritus John Marsh Cancer Center, Hagerstown, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Reliant Medical Group, Inc., Worcester, Massachusetts
  - Mayo Clinic in Rochester, Minnesota, Rochester, Minnesota
  - Jackson Oncology Associates PLLC, Jackson, Mississippi
  - HCA Midwest Kansas City, MidAmerica Division, Inc., Kansas City, Missouri
  - Cancer Alliance of Nebraska, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Tennessee Cancer Specialists, Omaha, Nebraska
  - Renown Regional Medical Center, Reno, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering - Basking Ridge, Basking Ridge, New Jersey
  - Summit Medical Group Cancer Center, Florham Park, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - The Valley Hospital, Inc., Paramus, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Broome Oncology, Binghamton, New York
  - Weill Cornell Medical College, New York, New York
  - Vassar Brothers Medical Center, Poughkeepsie, New York
  - SUNY At Stony Brook, Stony Brook, New York
  - White Plains Hospital, White Plains, New York
  - WakeMed Cancer Care - Waverly Hematology & Medical Oncology, Cary, North Carolina
  - Margaret R. Pardee Memorial Hospital, Hendersonville, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Aultman Hospital, Canton, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Columbus Community Clinical Oncology Program, Columbus, Ohio
  - Asante Rogue Regional Medical Center, Medford, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Abington Medical Specialists, Abington, Pennsylvania
  - St. Luke's Hospital & Health Network, Bethlehem, Pennsylvania
  - Albert Einstein Healthcare Network, Philadelphia, Pennsylvania
  - AHN Allegheny General Hospital, Pittsburgh, Pennsylvania
  - NSABP Foundation, Pittsburgh, Pennsylvania
  - PinnacleHealth Cancer Institute, Pittsburgh, Pennsylvania
  - Univ of Pittsburgh Cancer Inst. (UPCI), Pittsburgh, Pennsylvania
  - WellSpan Health/York Cancer Center Oncology Research, York, Pennsylvania
  - McLeod Regional Medical Center, Florence, South Carolina
  - St Francis Cancer Center, Greenville, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Sanford USD Medical Center, Sioux Falls, South Dakota
  - Erlanger Health System, Chattanooga, Tennessee
  - Chattanooga Research and Medicine, Chattanooga, Tennessee
  - The West Clinic, PLLC dba West Cancer Center, Germantown, Tennessee
  - Urology Associates of Kingsport, Kingsport, Tennessee
  - Tennessee Cancer Specialists, Knoxville, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - Baptist Cancer Center, Memphis, Tennessee
  - Florida Cancer Specialists, Nashville, Tennessee
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Tennessee Oncology Nashville, Nashville, Tennessee
  - Texas Oncology Cancer Care and Research Center, Austin, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - Texas Oncology Fort Worth, Fort Worth, Texas
  - Oncology Consultants, P.A., Houston, Texas
  - Texas Oncology P.A., Lewisville, Texas
  - University of Texas Health Science Center - San Antonio, San Antonio, Texas
  - Arizona Oncology Associates, P.C. - HOPE, The Woodlands, Texas
  - Comprehensive Cancer Centers of Nevada, The Woodlands, Texas
  - Illinois Cancer Specialists, The Woodlands, Texas
  - Miami Cancer Institute at Baptist Health, Inc., The Woodlands, Texas
  - Minnesota Oncology/Hematology PA, The Woodlands, Texas
  - Northwest Cancer Specialists PC, The Woodlands, Texas
  - Oncology and Hematology Associates of Southwest Virginia Inc, The Woodlands, Texas
  - Oncology Hematology Care Inc, The Woodlands, Texas
  - Oncology Hematology West, The Woodlands, Texas
  - Sansum Clinic, The Woodlands, Texas
  - Shenandoah Oncology, P.C., The Woodlands, Texas
  - Texas Oncology - Dallas Presbyterian Hospital, The Woodlands, Texas
  - Texas Oncology - Denison, The Woodlands, Texas
  - Texas Oncology - McAllen, The Woodlands, Texas
  - Texas Oncology - McKinney, The Woodlands, Texas
  - Texas Oncology - Medical City Dallas, The Woodlands, Texas
  - Texas Oncology - Methodist Dallas Cancer Center, The Woodlands, Texas
  - Texas Oncology - Paris, The Woodlands, Texas
  - Texas Oncology - San Antonio Medical Center, The Woodlands, Texas
  - Texas Oncology - The Woodlands, The Woodlands, Texas
  - Texas Oncology - Tyler, The Woodlands, Texas
  - Texas Oncology - West Texas, The Woodlands, Texas
  - Texas Oncology Cancer Care and Research Center, The Woodlands, Texas
  - Texas Oncology Denton, The Woodlands, Texas
  - Texas Oncology Fort Worth, The Woodlands, Texas
  - Texas Oncology P.A., The Woodlands, Texas
  - Texas Oncology- Mesquite, The Woodlands, Texas
  - Texas Oncology-Arlington South, The Woodlands, Texas
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, The Woodlands, Texas
  - Texas Oncology-Deke Slayton Cancer Center, The Woodlands, Texas
  - Texas Oncology-Plano East, The Woodlands, Texas
  - Texas Oncology-Plano West, The Woodlands, Texas
  - US Oncology, The Woodlands, Texas
  - USO - Texas Oncology, P. A., The Woodlands, Texas
  - USO-Maryland Oncology Hematology, P.A., The Woodlands, Texas
  - USO-New York Oncology Hematology, P.C, The Woodlands, Texas
  - USO-Rocky Mountain Cancer Center, The Woodlands, Texas
  - USO-Southern Cancer Center, P.C., The Woodlands, Texas
  - USO-Virginia Oncology Associates, The Woodlands, Texas
  - Virginia Cancer Specialists, The Woodlands, Texas
  - Willamette Valley Cancer Institute & Research Ctr., The Woodlands, Texas
  - Texas Oncology - Paris, Tyler, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - The University of Vermont Medical Center Inc., Burlington, Vermont
  - Hematology Oncology Associates of Fredericksburg Inc., Fredericksburg, Virginia
  - Virginia Commonwealth University (VCU) Medical Center, Richmond, Virginia
  - MultiCare Regional Cancer Center - Auburn, Auburn, Washington
  - Swedish Medical Center, Seattle, Washington
- Argentina (15):
  - Centro de Oncologia e Investigacion Buenos Aires, Berazategui, Buenos Aires
  - Instituto de Investigaciones Clinicas Mar del Plata, Mar del Plata, Buenos Aires
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Hospital Aleman, Buenos Aires, Buenos Aires F.D.
  - Fundacion CENIT para la Investigacion en Neurociencias, CABA, Ciudad Autonoma Buenos Aires
  - Clinica Viedma, Viedma, Río Negro Province
  - Instituto de Oncologia de Rosario, Rosario, Santa Fe Province
  - Centro Para la Atención Integral del Paciente Oncologico (CAIPO), San Miguel de Tucumán, Tucumán Province
  - Instituto Alexander Fleming, Buenos Aires
  - IDIM - Instituto de Diagnóstico e Investigaciones Metabólicas, Buenos Aires
  - Clinica Adventista de Belgrano, Ciudad Autonoma Buenos Aires
  - Fundación CORI para la Investigación y Prevención del Cáncer, La Rioja
  - Consultorio Dr. Miguel Ángel Escudero, Salta
  - CER San Juan, San Juan
  - Centro Medico San Roque, San Miguel de Tucumán
- Australia (20):
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - St Vincent's Hospital, Darlinghurst, New South Wales
  - Lismore Base Hospital, Lismore, New South Wales
  - Liverpool Hospital, Liverpool, New South Wales
  - Mater Hospital Sydney, Sydney, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Southern Medical Day Care Centre, Wollongong, New South Wales
  - Mater Misericordiae Limited, Brisbane, Queensland
  - Gold Coast University Hospital, Southport, Queensland
  - The Townsville Hospital, Townsville, Queensland
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Ashford Cancer Centre Research, Kurralta Park, South Australia
  - Launceston General Hospital, Launceston, Tasmania
  - Box Hill Hospital, Box Hill, Victoria
  - Epworth Hospital, East Melbourne, Victoria
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Maroondah Hospital, Melbourne, Victoria
  - Breast Cancer Research Centre WA, Nedlands, Western Australia
  - St John of God Subiaco Hospital, Subiaco, Western Australia
- Austria (7):
  - Medizinische Universität Graz, Graz, Styria
  - Medizinische Universitaet Innsbruck, Innsbruck, Tyrol
  - Private Practice - Dr. Hubalek, Schwaz, Tyrol
  - Medizinische Universität Wien, Vienna, Vienna
  - Universitaetsklinikum Allgemeines Krankenhaus Wien, Vienna, Vienna
  - Klinik Hietzing, Vienna, Vienna
  - Universitätsklinikum Salzburg, Salzburg
- Belgium (17):
  - Algemeen Ziekenhuis klina, Brasschaat, Antwerpen
  - Antwerp University Hospital, Edegem, Antwerpen
  - Cliniques Universitaires Saint-Luc, Brussels, Bruxelles-Capitale, Région de
  - CHU de Charleroi - Hopital Civil Marie Curie, Lodelinsart, Hainaut
  - Jessa Ziekenhuis, Hasselt, Limburg
  - Centre Hospitalier Universitaire de Liège - Domaine Universitaire du Sart Tilman, Liège, Liège
  - Centre Hospitalier D'Ardenne - Forget, Libramont, Luxembourg
  - Université Catholique de Louvain-Namur - Centre Hospitalier Universitaire Dinant-Godinne - Site Godinne, Yvoir, Namur
  - AZ Nikolaas, Sint-Niklaas, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams-Brabant
  - Groupe Jolimont, La Louvière, Wallonne, Région
  - Clinical Chc Montlégia, Liège, Wallonne, Région
  - Clinique Saint Pierre, Ottignies, Wallonne, Région
  - AZ Sint-Jan Brugge-Oostende AV, Bruges, West-Vlaanderen
  - Jan Yperman ziekenhuis, Ieper, West-Vlaanderen
  - AZ Groeninge Campus Kennedylaan, Kortrijk, West-Vlaanderen
  - CHU UCL Namur/Site Sainte Elisabeth, Namur
- Brazil (20):
  - Centro de Pesquisa Clínica do Instituto do Câncer do Ceará, Fortaleza, Ceará
  - Sírio-Libanês Brasilia-Centro de Oncologia-Asa Sul, Brasília, Federal District
  - Hospital Araújo Jorge, Goiânia, Goiás
  - CIONC - Centro Integrado de Oncologia de Curitiba, Curitiba, Paraná
  - Hospital de Cancer de Londrina, Londrina, Paraná
  - Instituto de Educação, Pesquisa e Gestão em Saúde, Rio de Janeiro, Rio de Janeiro
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia, Ijuí, Rio Grande do Sul
  - Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Hospital de Clínicas de Ribeirão Preto, Ribeirão Preto, São Paulo
  - Faculdade de Medicina do ABC, Santo André, São Paulo
  - Hospital de Base de São José do Rio Preto, Sao Jose Rio Preto, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - INCA - Instituto Nacional Do Cancer, Rio de Janeiro
  - Hospital Sírio Libanês, São Paulo
  - Pérola Centro de Pesquisa em Oncologia, São Paulo
  - IBCC - Núcleo de Pesquisa e Ensino, São Paulo
  - Instituto de Assistência Médica ao Servidor Público Estadual - IAMSPE/HSPE-FMO Conhecer Centro de Oncolog -T, São Paulo
  - Instituto D'Or de Pesquisa e Ensino (IDOR), São Paulo
- Canada (9):
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - North York General Hospital, Toronto, Ontario
  - Humber River Hospital, Toronto, Ontario
  - Unity Health Toronto, St. Michael's Hospital, Toronto, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
  - CHU de Quebec-Hopital de Saint-Sacrement, Québec, Quebec
  - Centre intégré universitaire de santé et de services sociaux de l'Estrie - Centre Hospitalier Universitair -T, Sherbrooke, Quebec
- China (16):
  - The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Fujian Medical University Union Hospital-1 Bingfanglou, Fuzhou, Fujian
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun-Yat Sen University, Guangzhou, Guangdong
  - Sun Yat-Sen University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital, Nanjing, Nanjing
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai Jiaotong University School of Medicine Ruijin Hospital, Shanghai, Shanghai Municipality
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Czechia (6):
  - Nemocnice Horovice, Hořovice, Beroun
  - Masarykuv onkologicky ustav, Brno, Brno-město
  - Fakultni Nemocnice Ostrava, Ostrava, Moravskoslezský kraj
  - Multiscan, Pardubice, Pardubický kraj
  - Fakultni Thomayerova nemocnice, Prague, Praha 4
  - FN Plzen Lochotin, Pilsen
- Denmark (10):
  - Herlev and Gentofte Hospital, Copenhagen, Capital Region
  - Rigshospitalet, København Ø, Capital Region
  - Aarhus Universitetshospital, Skejby, Aarhus, Central Jutland
  - Regionshospitalet Herning, Herning, Central Jutland
  - Aalborg Universitetshospital, Syd, Aalborg, North Denmark
  - Næstved Sygehus, Næstved, Region Sjælland
  - Sydvestjysk Sygehus Esbjerg, Esbjerg, Region Syddanmark
  - Odense Universitetshospital, Odense, Region Syddanmark
  - Sygehus Soenderjylland, Sønderborg, Region Syddanmark
  - Vejle Sygehus, Vejle, Region Syddanmark
- Finland (9):
  - Keski-Suomen Keskussairaala, Jyväskylä, Central Finland
  - Oulun yliopistollinen sairaala, Oulu, North Ostrobothnia
  - Kuopion Yliopistollinen Sairaala, Kuopio, Northern Savonia
  - Tampereen yliopistollinen sairaala, Tampere, Pirkanmaa
  - Vaasan Keskussairaala, Vaasa, Pohjanmaa
  - Satakunnan Keskussairaala, Pori, Satakunta
  - Turku University Central Hospital, Turku, Southwest Finland
  - Docrates Syöpäsairaala, Helsinki, Uusimaa
  - Päijät-Häme Central hospital, Lahti
- France (17):
  - Centre Leon Berard, Lyon, Auvergne-Rhône-Alpes
  - Centre Hospitalier Régional Universitaire de Brest - Hôpital Morvan, Brest, Brittany Region
  - Polyclinique De Blois, La Chaussée-Saint-Victor, Centre-Val de Loire
  - Centre Georges Francois Leclerc, Dijon, Côte-d'Or
  - Hôpital Privé des Côtes d'Armor- HPCA, Plérin, Côtes-d'Armor
  - CHU de Besancon Hopital Jean Minjoz, Besançon, Doubs
  - Centre Eugène Marquis Rennes - Centre de Lutte Contre le Cancer, Rennes, Ille-et-Vilaine
  - Centre de Cancérologie du Grand Montpellier, Montpellier, Languedoc-Roussillon
  - Institut de Cancérologie de l'Ouest, Saint-Herblain, Loire-Atlantique
  - Polyclinique de Gentilly, Nancy, Meurthe-et-Moselle
  - Clinique Victor Hugo Le Mans, Le Mans, Pays de la Loire Region
  - Centre Jean Perrin - Centre Régional de Lutte contre le Cancer d'Auvergne, Clermont-Ferrand, Puy-de-Dôme
  - Henri Mondor Hospital, Créteil, Seine-et-Marne
  - Centre de Lutte Contre le Cancer - Centre Henri Becquerel Normandie Rouen, Rouen, Seine-Maritime
  - Sainte Catherine Institut du Cancer Avignon Provence, Avignon, Vaucluse
  - Centre Hospitalier de Vendee Les Oudairies, La Roche-sur-Yon, Vendée
  - Institut Curie, Paris
- Germany (33):
  - Praxis für interdisziplinäre Onkologie & Hämatologie, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Private Practice - Dr. Helmut Oettle und Prof.Dr.med. Frank Mayer, Friedrichshafen, Baden-Wurttemberg
  - Klinikum Ludwigsburg, Ludwigsburg, Baden-Wurttemberg
  - Universitätsklinikum Tübingen, Tübingen, Baden-Wurttemberg
  - Universitätsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Klinikum St. Marien Amberg, Amberg, Bavaria
  - Gemeinschaftspraxis hop-augsburg, Augsburg, Bavaria
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Klinikum der Ludwig-Maximilians-Universitaet Muenchen, München, Bavaria
  - Klinikum Rechts Der Isar Der Technischen Universität München, München, Bavaria
  - Rotkreuzklinikum München gemeinnützige GmbH, München, Bavaria
  - Agaplesion Markus Krankenhaus, Frankfurt am Main, Hesse
  - Private Practice - Dres. Andreas Köhler und Roswitha Fuchs, Langen, Hesse
  - Sana Klinikum Offenbach, Offenbach, Hesse
  - Franziskus-Hospital Harderberg, Georgsmarienhütte, Lower Saxony
  - Gynäkologisch-Onkologische Praxis am Pelikanplatz, Hanover, Lower Saxony
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Universitätsklinikum Bonn, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Düsseldorf, Düsseldorf, North Rhine-Westphalia
  - Kliniken Essen-Mitte, Evangelische Huyssens-Stiftung, Essen, North Rhine-Westphalia
  - Zentrum fuer ambulante gynaekologische Onkologie (ZAGO), Krefeld, North Rhine-Westphalia
  - Evangelisches Krankenhaus Bethesda Mönchengladbach gGmbH, Mönchengladbach, North Rhine-Westphalia
  - Universitätsklinikum Münster - Albert Schweitzer Campus, Münster, North Rhine-Westphalia
  - Marien Hospital Witten, Witten, North Rhine-Westphalia
  - Universitätsklinikum Carl Gustav Carus, Dresden, Saxony
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel, Kiel, Schleswig-Holstein
  - SRH Wald-Klinikum Gera gGmbH, Gera, Thuringia
  - Helios Klinikum Berlin-Buch, Berlin
  - Medizinisches Versorgungszentrum Onkologischer Schwerpunkt am Oskar-Helene-Heim, Berlin
  - Mammazentrum HH - Krankenhaus Jerusalem, Hamburg
  - Kath. Marienkrankenhaus gGmbH, Hamburg
  - Asklepios Kliniken Hamburg, Hamburg
- Greece (13):
  - University Hospital of Patras, Pátrai, Achaia
  - Errikos Dunant Hospital Center, Athens, Attikí (Region)
  - Alexandra Hospital, Athens, Attikí
  - Agios Savvas Regional Cancer Hospital, Athens, Attikí
  - Metropolitan Hospital, Athens, Attikí
  - Attikon General University Hospital, Chaïdári, Attikí
  - General Oncology Hospital of Kifissia "Agioi Anargiroi", Nea Kifissia, Attikí
  - Bioclinic of Thessaloniki, Thessaloniki, Kentrikí Makedonía
  - University General Hospital of Heraklion, Heraklion, Krítí
  - European Interbalkan Medical Center, Thessaloniki, Thessaloníki
  - Euromedica - General Clinic of Thessaloniki, Thessaloniki
  - Papageorgiou General Hospital of Thessaloniki, Thessaloniki
  - University Hospital of Ioannina, Ioannina, Ípeiros
- Hong Kong (4):
  - Pamela Youde Nethersole Eastern Hospital, Chai Wan
  - Queen Mary Hospital, Hksar
  - Tuen Mun Hospital, Tuenmen
  - Queen Elizabeth Hospital, Yau Ma Tei
- Hungary (7):
  - Bacs-Kiskun Varmegyei Oktatokorhaz, Kecskemét, Bács-Kiskun county
  - Jasz-Nagykun-Szolnok Megyei Hetenyi Geza Korhaz, Szolnok, Jász-Nagykun-Szolnok
  - Szent Margit Kórház, Budapest
  - Magyar Honvedseg Egeszsegugyi Kozpont, Budapest
  - Semmelweis University, Budapest
  - Szent Imre Egyetemi Oktatokorhaz, Budapest
  - Uzsoki Utcai Kórház, Budapest
- India (15):
  - MNJ Institute of Oncology, Hyderabad, Andhra Pradesh
  - HCG Cancer Centre, Ahmedabad, Gujarat
  - HCG Cancer Centre, Vadodara, Gujarat
  - Artemis Hospital, Gurgaon, Haryana
  - Manipal Hospital, Bangalore, Karmnataka
  - Regional Cancer Centre, Trivandrum, Kerala
  - Tata Memorial Hospital, Mumbai, Maharashtra
  - HCG Manavata Cancer Centre, Nashik, Maharashtra
  - Grant Medical Foundation - Ruby Hall Clinic, Pune, Maharashtra
  - Deenanth Mangeshkar Hospital and Research Centre, Pune, Maharashtra
  - Dr. B. L. Kapur Memorial Hospital, New Delhi, National Capital Territory of Delhi
  - Apollo Speciality Hospital - Teynampet, Chennai, Tamil Nadu
  - Apollo Gleneagles Hospitals, Kolkata, West Bengal
  - Medica Superspecialty Hospital, Kolkata, West Bengal
  - Post Graduate Institute of Medical Education & Research, Chandigarh
- Israel (9):
  - Meir Medical Center, Kfar Saba, Central District
  - Rabin Medical Center, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Kaplan Medical Center, Rehovot, Central District
  - Yitzhak Shamir Medical Center, Ẕerifin, Central District
  - Shaare Zedek Medical Center, Jerusalem, Jerusalem
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Soroka Medical Center, Beersheba, Southern District
  - Rambam Health Care Campus, Haifa, Ḥeifā
- Italy (18):
  - University of Naples Federico II, Napoli, Campania
  - Azienda Ospedaliero Universitaria S.Anna, Cona, Emilia-Romagna
  - Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori, Meldola, Emilia-Romagna
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Lombardy
  - Ospedale Fatebenefratelli-Oftalmico, Milan, Milano
  - Humanitas, Rozzano, Milano
  - Istituto Nazionale Tumori Regina Elena, Rome, Roma
  - Azienda Ospedaliera Sant'Andrea, Rome, Roma
  - Azienda Ospedaliera Santa Maria, Terni, TR
  - Ospedale Bellaria - Azienda USL di Bologna, Bologna
  - Ospedale Antonio Perrino, Brindisi
  - Ospedale San Martino, Genova
  - Azienda Ospedaliero Universitaria, Modena
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli
  - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliera Di Parma, Parma
  - Azienda Ospedaliero-Universitaria Città della Salute e della Scienza di Torino, Torino
  - APSS - Presidio Ospedaliero Santa Chiara, Trento
- Japan (35):
  - Aichi Cancer Center Hospital, Nagoya, Aichi-ken
  - Chiba Cancer Center, Chiba, Chiba
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Kurume General Hospital, Kurume, Fukuoka
  - Gunma Prefectural Cancer Center, Ōta, Gunma
  - Hiroshima University Hospital, Hiroshima, Hiroshima
  - National Hospital Organization Hokkaido Cancer Center, Sapporo, Hokkaido
  - Hyogo College of Medecine, Nishinomiya, Hyōgo
  - University of tsukuba hospital, Tsukuba, Ibaragi
  - Tokai University Hospital- Isehara Campus, Isehara, Kanagawa
  - St Marianna University School of Medicine Hospital, Kawasaki, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - KKR Tohoku Kosai Hospital, Aoba-ku, Sendai-shi, Miyagi
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Kindai University Hospital- Osakasayama Campus, Osaka Sayama-shi, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Saitama Prefectural Cancer Center, Ina-machi, Saitama
  - Shizuoka Cancer Center, Nakatogari, Shizuoka
  - Jichi Medical University Hospital, Shimotsuke, Tochigi
  - Tochigi Cancer Center, Utsunomiya, Tochigi
  - Juntendo University Hospital, Bunkyō-Ku, Tokyo
  - National Cancer Center Hospital, Chuo Ku, Tokyo
  - St. Lukes International Hospital, Chuo-Ku, Tokyo
  - Japanese Foundation for Cancer Research, Koto, Tokyo
  - Showa University Hospital, Shinagawa-ku, Tokyo
  - Tokyo Medical University Hospital, Shinjuku-ku, Tokyo
  - National Center for Global Health and Medicine, Shinjuku-ku, Tokyo
  - National Hospital Organization Kyushu Cancer Center, Fukuoka
  - Sagara Hospital, Kagoshima
  - Kumamoto University Hospital, Kumamoto
  - Kumamoto Shinto General hospital, Kumamoto
  - Kyoto University Hospital, Kyoto
  - National Hospital Organization Osaka Medical Center, Osaka
  - Osaka International Cancer Institute, Osaka
- Mexico (17):
  - CIMAB S.A. de C.V., Torreón, Coahuila
  - Health Pharma Professional Research, S.A. de C.V., Mexico City, Federal District
  - Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco
  - Centro Oncológico Internacional (COI), Guadalajara, Jalisco
  - Grupo Medico Camino S.C., Mexico City, Mexico City
  - Centro Regiomontano de Investigacion, Monterrey, Nuevo León
  - Private Practice - Dr. Joaquin Reinoso, Monterrey, Nuevo León
  - Filios Alta Medicina, Monterrey, Nuevo León
  - Centro de Estudios y Prevencion del Cancer, Juchitán de Zaragoza, Oaxaca
  - Neurociencias Estudios Clinicos S.C., Culiacán, Sinaloa
  - Centro Hemato Oncologico Privado, Toluca, Toluca
  - Medical Care and Research, S.A. de C.V., Mérida, Yucatán
  - Centro de Atención e Investigación Clínica en Oncología, Mérida, Yucatán
  - Unidad de Investigacion en Salud, Chihuahua City
  - Oaxaca Site Management Organization SC, Oaxaca City
  - Unidad Médica Onco-hematológica, Puebla City
  - Oncológico Potosino, San Luis Potosí City
- Netherlands (4):
  - Maastricht UMC+, Maastricht, Limburg
  - Onze Lieve Vrouwe Gasthuis (OLVG), Amsterdam, North Holland
  - Albert Schweitzer Ziekenhuis, locatie Dordwijk, Dordrecht, South Holland
  - Haga Ziekenhuis locatie Leyweg, The Hague, South Holland
- New Zealand (3):
  - Waikato Hospital, Hamilton, Waikato Region
  - Palmerston North Hospital, Palmerston North, Wanganui
  - Auckland City Hospital, Auckland
- Poland (11):
  - Przychodnia Lekarska "Komed", Konin, Greater Poland Voivodeship
  - Wielkopolskie Centrum Onkologii, Poznan, Greater Poland Voivodeship
  - Dolnośląskie Centrum Onkologii we Wrocławiu, Wroclaw, Lower Silesian Voivodeship
  - Centrum Onkologii Ziemii Lubelskiej, Lublin, Lublin Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie, Warsaw, Masovian Voivodeship
  - Luxmed Onkologia sp. z o. o., Warsaw, Masovian Voivodeship
  - Opolskie Centrum Onkologii w Opolu im. prof. Tadeusza Koszarowskiego, Opole, Opole Voivodeship
  - Uniwersyteckie Centrum Kliniczne, Gdansk, Pomeranian Voivodeship
  - Szpitale Pomorskie Sp. z o. o., Gdynia, Pomeranian Voivodeship
  - Olsztyński Ośrodek Onkologiczny Kopernik, Olsztyn, Warmian-Masurian Voivodeship
  - Centrum Terapii Wspolczesnej J. M. Jasnorzewska Spolka Komandytowo-Akcyjna, Lodz, Łódź Voivodeship
- Portugal (5):
  - Instituto Portugês de Oncologia de Coimbra Francisco Gentil, Coimbra
  - Champalimaud Foundation, Lisbon
  - Centro Hospitalar Lisboa Norte, E.P.E. - Hospital de Santa Maria, Lisbon
  - Centro Hospitalar do Porto - Hospital de Santo António, Porto
  - IPOFG - Porto, Porto
- Puerto Rico (2):
  - Puerto Rico Hematology/Oncology Group, Bayamón, PR
  - UPR Comprehensive Cancer Center, San Juan, PR
- Romania (7):
  - Institutul Oncologic, Bucharest, București
  - Institutul Oncologic, Cluj-Napoca, Cluj
  - Ovidius Clinical Hospital OCH, Ovidiu, Constanța County
  - Centrul de Oncologie "Sfântul Nectarie", Craiova, Dolj
  - Radiology Therapeutic Center, Otopeni, Ilfov
  - Oncopremium Team, Baia Mare, Maramureş
  - Spitalul Clinic Filantropia, Bucharest
- Russia (16):
  - Chelyabinsk Regional Oncology Dispensary, Chelyabinsk, Chelyabinsk Oblast
  - Kaluga Regional Clinical Oncology Center, Kaluga, Kalužskaja Oblast'
  - Kursk Regional Oncology Dispensary, Kursk, Kursk Oblast
  - Fed State Budgetary Inst "N.N. Blokhin Med Center of Oncology" MHRF, Moscow, Moscow
  - Burdenko Main Military Hospital, Moscow, Moscow
  - Orenburg Regional Clinical Oncology Dispensary, Orenburg, Orenburg Oblast
  - Samara Regional Clinical Oncology Center, Samara, Samara Oblast
  - Leningrad Regional Oncology Dispensary, Saint Petersburg, Sankt-Peterburg
  - North-Western State Medical University named after I.I.Mechnikov, Saint Petersburg, Sankt-Peterburg
  - St. Petersburg City Oncological Dispensary - Berezovaya Avenue, Saint Petersburg, Sankt-Peterburg
  - N.N.Petrov Research Institute of Oncology, Saint Petersburg, Sankt-Peterburg
  - Saint-Petersburg Scientific-Practical Center of Specialized Kinds of Medical Care (oncological) named afte -T, Saint Petersburg, Sankt-Peterburg
  - Republican Clinical Oncology Dispensary, Kazan', Tatarstan Republic
  - Volgograd Regional Oncological Dispensary No. 3, Volzhsky, Volgograd Oblast
  - Yaroslavl Regional Cancer Hospital, Yaroslavl, Yaroslavl Oblast
  - Blokhin Cancer Research Center, Moscow
- Saudi Arabia (4):
  - King Fahad Specialist Hospital-Dammam, Dammam, Eastern Province
  - King Abdulaziz Medical City - National Guard Hospital, Riyadh, Riyadh Region
  - King Fahad Medical City, Riyadh, Riyadh Region
  - King Faisal Specialist Hospital & Research Center, Riyadh
- Singapore (2):
  - National Cancer Center, Singapore, Central Singapore
  - National University Hospital, Singapore
- South Africa (6):
  - Cancercare Langenhoven Drive Oncology Centre, Port Elizabeth, Eastern Cape
  - Life Groenkloof, Pretoria, Gauteng
  - Eastleigh Breast Care Center, Pretoria, Gauteng
  - Sandton Oncology Medical Group (Pty) Ltd, Sandton, Gauteng
  - Cancercare Rondebosch Oncology, Cape Town, Western Cape
  - GVI Oncology, George, Western Cape
- South Korea (16):
  - Chungbuk National University Hospital, Cheongju-si, Chungcheongbuk-do [Chungbuk]
  - Soon chun hyang University Cheonan Hospital, Cheonan-si, Chungcheongnam-do [Chungnam]
  - Inha University Hospital, Incheon, Incheon-gwangyeoksi [Incheon]
  - Gachon University Gil Medical Center, Namdong-gu, Incheon-gwangyeoksi [Incheon]
  - National Cancer Center, Goyang-si, Kyǒnggi-do
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Dongnam Institute of Radiological and Medical Sciences, Busan, Pusan-Kwangyǒkshi
  - Inje University Haeundae Paik Hospital, Haeundae-gu, Pusan-Kwangyǒkshi
  - Korea University Anam Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Severance Hospital Yonsei University Health System, Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Korea University Guro Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Ewha Womans University Mokdong Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
  - Kyungpook National University Chilgok Hospital, Daegu, Taegu-Kwangyǒkshi
- Spain (28):
  - Hospital Universitario Reina Sofia, Córdoba, Andalusia
  - Hospital Quiron Barcelona, Barcelona, Barcelona [Barcelona]
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [Cataluña]
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalunya [Cataluña]
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, La Coruna
  - Hospital Universitario Arnau de Vilanova de Lleida, Lleida, Lleida [Lérida]
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid
  - Hospital Universitario Fundacion ALcorcon, Alcorcón, Madrid, Comunidad de
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital Universitario Virgen de la Victoria, Málaga, Málaga
  - Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital Clínico de Valencia, Valencia, Valenciana, Comunitat
  - Parc de Salut Mar - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario San Cecilio, Granada
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital La Princesa, Madrid
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario HM Sanchinarro, Madrid
  - Hospital Universitario de Salamanca - Complejo Asistencial Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitario Virgen de Valme, Seville
  - Hospital Quirón Salud Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Sweden (5):
  - Skånes universitetssjukhus Lund, Malmo, Skåne Län [se-12]
  - Norrlands universitetssjukhus, Umeå, Västerbottens Län [se-24]
  - Sundsvalls Sjukhus, Sundsvall, Västernorrlands Län [se-22]
  - Västmanlands sjukhus Västerås, Västerås, Västmanlands Län [se-19]
  - Växjö Centrallasarettet, Vaxjo
- Taiwan (11):
  - Chang Gung Memorial Hospital - Kaohsiung, Kaohsiung Niao Sung Dist, Kaohsiung
  - Tri-Service General Hospital, Taipei City, Taipei
  - Changhua Christian Hospital, Changhua
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taipei Medical University Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - MacKay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan
- Turkey (Türkiye) (14):
  - Istanbul Universitesi Cerrahpasa, Istanbul- Fatih, Istanbul
  - Acibadem Altunizade Hospital, Üsküdar/stanbul, Istanbul
  - Ege University Medicine of Faculty, Bornova, İzmir
  - Izmir Medical Park Hospital, Izmir, Karsiyaka, İzmir
  - Ankara Gülhane Eitim ve Aratrma Hastanesi, Ankara, Kecioren
  - Baskent University Dr. Turgut Noyan Research and Training Center, Adana
  - Ankara Universitesi Tip Fakultesi Hastanesi, Ankara
  - Abdurrahman Yurtaslan Ankara Oncology, education and Research Hospital, Ankara
  - Hacettepe Universitesi, Ankara
  - Akdeniz Universitesi Hastanesi, Antalya
  - Trakya University Faculty of Medicine, Edirne
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Kocaeli Üniversitesi, Kocaeli
  - İnönü Üniversitesi Turgut Özal Tıp Merkezi, Malatya
- Ukraine (7):
  - Municipal Non-profit Enterprise "City Clinical Hospital #4" of Dnipro City Council, Dnipro, Dnipropetrovsk Oblast
  - Communal Enterprise 'Kryvyi Rih Oncology Dispensary' of the Dnipropetrovsk Regional Council, Kryvyi Rih, Dnipropetrovsk Oblast
  - Municipal non-profit enterprise'Odesa Regional Clinical Hospital'of Odesa Regional Council, Odesa, Odesa Oblast
  - Poltava Regional Clinical Oncology Center, Poltava, Poltava Oblast
  - Communal Noncommercial Enterprise "Podillia Regional Oncology Center Of Vinnytsia Regional Council", Vinnytsia, Vinnytsia Oblast
  - Municipal Enterprise "Volyn Regional Medical Oncology Centre" of the Volyn Regional Council, Lutsk, Volyn Oblast
  - Uzhgorod Central City Clinical Hospital, Uzhhorod, Zakarpattia Oblast
- United Kingdom (19):
  - The Royal Cornwall Hospital, Truro, England
  - Mid Essex Hospital Services NHS Trust, Chelmsford, Essex
  - North Middlesex Hospital, London, Greater London
  - Charing Cross Hospital, London, Hammersmith and Fulham
  - Mount Vernon Hospital, Northwood, Hertfordshire
  - Victoria Hospital, Blackpool, Lancashire
  - Royal Preston Hospital, Preston, Lancashire
  - Boston Pilgrim Hospital, Boston, Lincolnshire
  - Sarah Canon Research Institute UK, London, London, City of
  - Guy's & St Thomas' NHS Foundation Trust, London, London, City of
  - James Cook University Hospital, Central Middlesbrough, Middlesbrough
  - Western General Hospital, Edinburgh, Midlothian
  - Nottingham City Hospital, Nottingham, Nottinghamshire
  - The Churchill Hospital, Oxford, Oxfordshire
  - Musgrove Park Hospital, Taunton, Somerset
  - Royal Surrey County Hospital, Guildford, Surrey
  - Royal Marsden Hospital, London, Sutton
  - Airedale General Hospital, Bradford
  - The Christie, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Derived] Zhang Q, Shen K, Song CG, Ouyang Q, Liu Z, Liu Q, Feng J, Chiu JWY, Tang J, Jiang Z, Tseng LM, Wang X, Yang L, Qian C, Shao Z. Abemaciclib combined with endocrine therapy as adjuvant treatment for hormone-receptor-positive, HER2-, high-risk early breast cancer: 5-year Chinese population analysis of the phase III randomized monarchE study. Ther Adv Med Oncol. 2024 Oct 23;16:17588359241286775. doi: 10.1177/17588359241286775. eCollection 2024. PMID 39463748
- [Derived] Johnston SRD, Rugo HS, Tolaney SM, Munoz Fernandez M, Wei R, Martin M. Abemaciclib plus endocrine therapy for HR+, HER2-, node-positive, high-risk early breast cancer: a plain language summary of the monarchE study. Future Oncol. 2024;20(28):2037-2048. doi: 10.1080/14796694.2024.2362095. Epub 2024 Jul 18. PMID 39023253
- [Derived] Rastogi P, O'Shaughnessy J, Martin M, Boyle F, Cortes J, Rugo HS, Goetz MP, Hamilton EP, Huang CS, Senkus E, Tryakin A, Cicin I, Testa L, Neven P, Huober J, Shao Z, Wei R, Andre V, Munoz M, San Antonio B, Shahir A, Harbeck N, Johnston S. Adjuvant Abemaciclib Plus Endocrine Therapy for Hormone Receptor-Positive, Human Epidermal Growth Factor Receptor 2-Negative, High-Risk Early Breast Cancer: Results From a Preplanned monarchE Overall Survival Interim Analysis, Including 5-Year Efficacy Outcomes. J Clin Oncol. 2024 Mar 20;42(9):987-993. doi: 10.1200/JCO.23.01994. Epub 2024 Jan 9. PMID 38194616
- [Derived] Johnston SRD, Toi M, O'Shaughnessy J, Rastogi P, Campone M, Neven P, Huang CS, Huober J, Jaliffe GG, Cicin I, Tolaney SM, Goetz MP, Rugo HS, Senkus E, Testa L, Del Mastro L, Shimizu C, Wei R, Shahir A, Munoz M, San Antonio B, Andre V, Harbeck N, Martin M; monarchE Committee Members. Abemaciclib plus endocrine therapy for hormone receptor-positive, HER2-negative, node-positive, high-risk early breast cancer (monarchE): results from a preplanned interim analysis of a randomised, open-label, phase 3 trial. Lancet Oncol. 2023 Jan;24(1):77-90. doi: 10.1016/S1470-2045(22)00694-5. Epub 2022 Dec 6. PMID 36493792
- [Derived] Toi M, Boyle F, Im YH, Reinisch M, Molthrop D, Jiang Z, Wei R, Sapunar F, Grimes BR, Nabinger SC, Johnston SRD. Adjuvant Abemaciclib Combined with Endocrine Therapy: Efficacy Results in monarchE Cohort 1. Oncologist. 2023 Jan 18;28(1):e77-e81. doi: 10.1093/oncolo/oyac234. PMID 36342342
- [Derived] Martin M, Hegg R, Kim SB, Schenker M, Grecea D, Garcia-Saenz JA, Papazisis K, Ouyang Q, Lacko A, Oksuzoglu B, Reeves J, Okera M, Testa L, Shimizu C, Denduluri N, Adamchuk H, Dakhil S, Wei R, Forrester T, Fernandez MM, Zimmermann A, Headley D, Johnston SRD. Treatment With Adjuvant Abemaciclib Plus Endocrine Therapy in Patients With High-risk Early Breast Cancer Who Received Neoadjuvant Chemotherapy: A Prespecified Analysis of the monarchE Randomized Clinical Trial. JAMA Oncol. 2022 Aug 1;8(8):1190-1194. doi: 10.1001/jamaoncol.2022.1488. PMID 35653145
- [Derived] Perachino M, Poggio F, Arecco L, Blondeaux E, Spinaci S, Marrocco C, Levaggi A, Lambertini M. Update on Pregnancy Following Breast Cancer Diagnosis and Treatment. Cancer J. 2022 May-Jun 01;28(3):176-182. doi: 10.1097/PPO.0000000000000599. PMID 35594464
- [Derived] Polewski MD, Nielsen GB, Gu Y, Weaver AT, Gegg G, Tabuena-Frolli S, Cajaiba M, Hanks D, Method M, Press MF, Gottstein C, Gruver AM. A Standardized Investigational Ki-67 Immunohistochemistry Assay Used to Assess High-Risk Early Breast Cancer Patients in the monarchE Phase 3 Clinical Study Identifies a Population With Greater Risk of Disease Recurrence When Treated With Endocrine Therapy Alone. Appl Immunohistochem Mol Morphol. 2022 Apr 1;30(4):237-245. doi: 10.1097/PAI.0000000000001009. PMID 35384873
- [Derived] Rugo HS, O'Shaughnessy J, Boyle F, Toi M, Broom R, Blancas I, Gumus M, Yamashita T, Im YH, Rastogi P, Zagouri F, Song C, Campone M, San Antonio B, Shahir A, Hulstijn M, Brown J, Zimmermann A, Wei R, Johnston SRD, Reinisch M, Tolaney SM; monarchE Committee Members. Adjuvant abemaciclib combined with endocrine therapy for high-risk early breast cancer: safety and patient-reported outcomes from the monarchE study. Ann Oncol. 2022 Jun;33(6):616-627. doi: 10.1016/j.annonc.2022.03.006. Epub 2022 Mar 23. PMID 35337972
- [Derived] Royce M, Osgood C, Mulkey F, Bloomquist E, Pierce WF, Roy A, Kalavar S, Ghosh S, Philip R, Rizvi F, Mixter BD, Tang S, Pazdur R, Beaver JA, Amiri-Kordestani L. FDA Approval Summary: Abemaciclib With Endocrine Therapy for High-Risk Early Breast Cancer. J Clin Oncol. 2022 Apr 10;40(11):1155-1162. doi: 10.1200/JCO.21.02742. Epub 2022 Jan 27. PMID 35084948
- [Derived] Johnston SRD, Harbeck N, Hegg R, Toi M, Martin M, Shao ZM, Zhang QY, Martinez Rodriguez JL, Campone M, Hamilton E, Sohn J, Guarneri V, Okada M, Boyle F, Neven P, Cortes J, Huober J, Wardley A, Tolaney SM, Cicin I, Smith IC, Frenzel M, Headley D, Wei R, San Antonio B, Hulstijn M, Cox J, O'Shaughnessy J, Rastogi P; monarchE Committee Members and Investigators. Abemaciclib Combined With Endocrine Therapy for the Adjuvant Treatment of HR+, HER2-, Node-Positive, High-Risk, Early Breast Cancer (monarchE). J Clin Oncol. 2020 Dec 1;38(34):3987-3998. doi: 10.1200/JCO.20.02514. Epub 2020 Sep 20. PMID 32954927
- See also: A Study to Compare Treatment After Surgery of Abemaciclib (LY2835219) Combined With Standard Endocrine Therapy Versus Endocrine Therapy Alone in Participants With Breast Cancer (monarchE) — https://trials.lillytrialguide.com/en-US/trial/3qEzEekhpuCEESS2KeSM8m

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Completers included participants who had recurrence disease, death due to any cause, and participants off treatment but on study follow-up.
Period: Overall Study
Arm/Group | 150 mg Abemaciclib + Endocrine Therapy | Endocrine Therapy
Started | 2808 | 2829
Received at Least One Dose of Study Drug | 2791 | 2800
Completed | 650 | 607
Not Completed | 2158 | 2222
Not completed — Withdrawal by Subject | 119 | 134
Not completed — Lost to Follow-up | 12 | 13
Not completed — Missing disposition data | 0 | 1
Not completed — On study treatment | 2027 | 2074

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- 150 mg Abemaciclib + Endocrine Therapy: Participants received Abemaciclib orally at 150 milligrams (mg) twice daily with at least 6 hours between doses for up to for up to 2 years or until evidence of disease recurrence or other discontinuation criteria were met, whichever occurs first. Endocrine therapy (physicians' choice) standard-of-care was administered according to package label until discontinuation criteria were met.
- Total: Total of all reporting groups
Arm/Group | 150 mg Abemaciclib + Endocrine Therapy | Endocrine Therapy | Total
Number analyzed (Participants) | 2808 | 2829 | 5637
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.20 (11.26) | 52.10 (11.20) | 52.10 (11.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2787 | 2814 | 5601
  Male | 21 | 15 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 355 | 378 | 733
  Not Hispanic or Latino | 1734 | 1738 | 3472
  Unknown or Not Reported | 719 | 713 | 1432
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 64 | 58 | 122
  Asian | 675 | 669 | 1344
  Native Hawaiian or Other Pacific Islander | 3 | 4 | 7
  Black or African American | 57 | 53 | 110
  White | 1947 | 1978 | 3925
  More than one race | 22 | 25 | 47
  Unknown or Not Reported | 40 | 42 | 82
Region of Enrollment [Count of Participants; unit: Participants]
  Argentina | 77 | 68 | 145
  Australia | 108 | 109 | 217
  Austria | 22 | 20 | 42
  Belgium | 65 | 51 | 116
  Brazil | 144 | 153 | 297
  Canada | 28 | 16 | 44
  China | 187 | 170 | 357
  Czechia | 15 | 12 | 27
  Denmark | 54 | 58 | 112
  Finland | 45 | 49 | 94
  France | 86 | 101 | 187
  Germany | 148 | 152 | 300
  Greece | 74 | 64 | 138
  Hong Kong | 8 | 12 | 20
  Hungary | 24 | 28 | 52
  India | 59 | 53 | 112
  Israel | 39 | 38 | 77
  Italy | 72 | 59 | 131
  Japan | 181 | 196 | 377
  Mexico | 104 | 121 | 225
  Netherlands | 5 | 14 | 19
  New Zealand | 21 | 22 | 43
  Poland | 65 | 60 | 125
  Portugal | 21 | 16 | 37
  Puerto Rico | 1 | 3 | 4
  Romania | 53 | 60 | 113
  Russia | 66 | 73 | 139
  Saudi Arabia | 5 | 9 | 14
  Singapore | 11 | 21 | 32
  South Africa | 3 | 6 | 9
  South Korea | 122 | 123 | 245
  Spain | 144 | 148 | 292
  Sweden | 7 | 5 | 12
  Taiwan | 64 | 60 | 124
  Turkey | 125 | 110 | 235
  Ukraine | 54 | 51 | 105
  United Kingdom | 99 | 100 | 199
  United States | 402 | 418 | 820

OUTCOME MEASURES:

1. Primary Outcome: Invasive Disease Free Survival (IDFS)
Description: IDFS, as defined by the STEEP System, was measured from the date of randomization to the date of first occurrence of one of the following events: ipsilateral invasive breast tumor recurrence, regional invasive breast cancer recurrence, distant recurrence, contralateral invasive breast cancer, second primary non-breast invasive cancer, death attributable to any cause.
Time Frame: Baseline to Recurrence or Death from Any Cause (Up to 32 Months)
Population: All randomized participants (including the censored participants). 2672 participants were censored in "150 mg Abemaciclib + Endocrine Therapy," 2642 participants were censored in "Endocrine Therapy."
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 150 mg Abemaciclib + Endocrine Therapy | Endocrine Therapy
Number analyzed (Participants) | 2808 | 2829
Months | NA [NA to NA] — There were not enough events to compute a median or 95% confidence interval. | NA [NA to NA] — There were not enough events to compute a median or 95% confidence interval.
Statistical Analysis 1: Comparison: 150 mg Abemaciclib + Endocrine Therapy vs Endocrine Therapy; Test type: Superiority; p = 0.00957, Log Rank; Stratified by Interactive Web Response Systems (IWRS) Geographical Region, IWRS Prior Treatment, IWRS Menopausal Status; Hazard Ratio (HR) = 0.747, 95% CI 2-sided [0.598 to 0.932] — Stratified by IWRS Geographical Region, IWRS Prior Treatment, IWRS Menopausal Status

2. Secondary Outcome: IDFS for Participants With Ki-67 Index ≥20%
Description: Outcome data will be provided after the study is completed.
Time Frame: Baseline to Recurrence or Death from Any Cause (Approximately 10 Years)
Reporting Status: Not Posted, anticipated posting 2029-06

3. Secondary Outcome: Distant Relapse-Free Survival (DRFS)
Description: Distant relapse-free survival is defined as the time from randomization to distant recurrence or death from any cause, whichever occurs first.
Time Frame: Baseline to Distant Recurrence or Death from Any Cause (Up to 32 Months)
Population: All randomized participants (including the censored participants). 2702 participants were censored in "150 mg Abemaciclib + Endocrine Therapy," 2677 participants were censored in "Endocrine Therapy."
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | 150 mg Abemaciclib + Endocrine Therapy | Endocrine Therapy
Number analyzed (Participants) | 2808 | 2829
Months | NA [NA to NA] — There were not enough events to compute a median or 95% confidence interval. | NA [NA to NA] — There were not enough events to compute a median or 95% confidence interval.
Statistical Analysis 1: Comparison: 150 mg Abemaciclib + Endocrine Therapy vs Endocrine Therapy; Test type: Superiority; Hazard Ratio (HR) = 0.717, 95% CI 2-sided [0.559 to 0.920] — Stratified by IWRS Geographical Region, IWRS Prior Treatment, IWRS Menopausal Status

4. Secondary Outcome: Overall Survival (OS)
Description: Outcome data will be provided after the study is completed.
Time Frame: Baseline to Death from Any Cause (Approximately 10 Years)
Reporting Status: Not Posted, anticipated posting 2029-06

5. Secondary Outcome: Pharmacokinetics (PK): Minimum Steady State Concentration (Cmin,ss) of Abemaciclib
Description: Pharmacokinetics (PK): Minimum Steady State Concentration (Cmin,ss) of Abemaciclib
Time Frame: Day 1 (2 hours post-dose), Days 30, 60, 90 post-dose
Population: All randomized participants who received at least one dose of Abemaciclib and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | 150 mg Abemaciclib + Endocrine Therapy
Number analyzed (Participants) | 483
Nanograms per milliliter (ng/mL) | 143 (110)

6. Secondary Outcome: Change From Baseline on the Functional Assessment of Cancer Therapy - Breast (FACT-B)
Description: Outcome data will be provided after the study is completed.
Time Frame: Baseline, Follow Up (Approximately 3 Years)
Reporting Status: Not Posted, anticipated posting 2029-06

7. Secondary Outcome: Change From Baseline on the Functional Assessment of Cancer Therapy - Endocrine Symptoms (FACT-ES)
Description: Outcome data will be provided after the study is completed.
Time Frame: Baseline, Follow Up (Approximately 3 Years)]
Reporting Status: Not Posted, anticipated posting 2029-06

8. Secondary Outcome: Change From Baseline on the Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F)
Description: Outcome data will be provided after the study is completed.
Time Frame: Baseline, Follow Up (Approximately 3 Years)]
Reporting Status: Not Posted, anticipated posting 2029-06

9. Secondary Outcome: Change From Baseline on the EuroQol Five-Dimension Five-Level Questionnaire (EQ-5D-5L)
Description: Outcome data will be provided after the study is completed.
Time Frame: Baseline, Follow Up (Approximately 3 Years)]
Reporting Status: Not Posted, anticipated posting 2029-06

ADVERSE EVENTS:
Time Frame: Baseline to 32 Months
Description: All randomized participants who received at least one dose of study drug. There are gender specific adverse events, occurring only in male or female participants. The number of participants exposed has been adjusted accordingly.
Arm/Group | 150 mg Abemaciclib + Endocrine Therapy | Endocrine Therapy
All-Cause Mortality (participants affected / at risk) | 38/2791 | 36/2800
Serious Adverse Events (participants affected / at risk) | 344/2791 | 202/2800
Other Adverse Events (participants affected / at risk) | 2723/2791 | 2318/2800
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 150 mg Abemaciclib + Endocrine Therapy (N=2791) | Endocrine Therapy (N=2800)
Anaemia (Blood and lymphatic system disorders) | 8 (8) | 2 (2)
Bone marrow oedema (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (5) | 1 (1)
Acute left ventricular failure (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 6 (6) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 4 (5) | 1 (1)
Cardiotoxicity (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 4 (4) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Angle closure glaucoma (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Eyelid ptosis (Eye disorders) | 1 (1) | 0 (0)
Macular hole (Eye disorders) | 1 (1) | 0 (0)
Macular pseudohole (Eye disorders) | 0 (0) | 1 (1)
Retinal detachment (Eye disorders) | 2 (2) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 3 (3) | 3 (3)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dental caries (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 15 (18) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastritis erosive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 2 (2)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 3 (4) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 6 (6) | 2 (2)
Pancreatitis acute (Gastrointestinal disorders) | 2 (2) | 0 (0)
Peritoneal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0)
Capsular contracture associated with breast implant (General disorders) | 2 (2) | 1 (2)
Chest pain (General disorders) | 4 (4) | 1 (1)
Fatigue (General disorders) | 2 (2) | 0 (0)
General physical health deterioration (General disorders) | 4 (4) | 0 (0)
Hyperplasia (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 2 (2) | 3 (3)
Inflammation (General disorders) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 2 (2)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 7 (7) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 10 (10) | 2 (2)
Cholecystitis acute (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 3 (3)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2) | 1 (1)
Jaundice (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 1 (1)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Abscess (Infections and infestations) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 3 (3) | 2 (2)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 1 (1)
Biliary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Breast abscess (Infections and infestations) | 3 (3) | 1 (1)
Breast cellulitis (Infections and infestations) | 5 (5) | 4 (4)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Campylobacter gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 11 (13) | 9 (9)
Cellulitis staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Clostridium colitis (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 1 (1) | 0 (0)
Coronavirus infection (Infections and infestations) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 2 (2)
Diverticulitis (Infections and infestations) | 3 (4) | 5 (5)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Erysipelas (Infections and infestations) | 5 (9) | 0 (0)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis clostridial (Infections and infestations) | 1 (1) | 0 (0)
Hepatitis e (Infections and infestations) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Infective pulmonary exacerbation of cystic fibrosis (Infections and infestations) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 7 (7) | 3 (3)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Lymphangitis (Infections and infestations) | 2 (2) | 0 (0)
Mastitis (Infections and infestations) | 3 (4) | 5 (5)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
Meningitis viral (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic infection (Infections and infestations) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 23 (23) | 14 (15)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia streptococcal (Infections and infestations) | 1 (1) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1) | 0 (0)
Postoperative wound infection (Infections and infestations) | 2 (2) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (2) | 2 (2)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (2)
Sepsis (Infections and infestations) | 5 (5) | 2 (2)
Septic shock (Infections and infestations) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 6 (6) | 0 (0)
Urinary tract infection (Infections and infestations) | 12 (12) | 4 (4)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Breast procedural complication (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Exposure during pregnancy (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Incisional hernia (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative adhesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Skin flap necrosis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 4 (4)
Wound necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 5 (5) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 5 (5) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1)
Occult blood (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 2 (2) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 7 (9) | 0 (0)
Food intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypovolaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metabolic acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Fistula (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/2770 (0) | 2/2785 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colorectal carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Endometrial neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/2770 (0) | 1/2785 (1)
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Meningioma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/2770 (1) | 2/2785 (2)
Carotid artery aneurysm (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 2 (2)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral infarction (Nervous system disorders) | 2 (2) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 1 (1)
Cerebral venous thrombosis (Nervous system disorders) | 2 (2) | 0 (0)
Cerebrospinal fluid leakage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 3 (3) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Monoparesis (Nervous system disorders) | 0 (0) | 1 (1)
Movement disorder (Nervous system disorders) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy (Nervous system disorders) | 1 (1) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 4 (4) | 2 (2)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 2 (2)
Trigeminal neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Device failure (Product Issues) | 0 (0) | 1 (1)
Bipolar disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1) | 1 (1)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Mania (Psychiatric disorders) | 0 (0) | 1 (1)
Mental disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 1 (1) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 4 (4) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 3 (3) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal impairment (Renal and urinary disorders) | 1 (1) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1)
Adenomyosis (Reproductive system and breast disorders) | 1/2770 (1) | 0/2785 (0)
Breast atrophy (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Breast calcifications (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast disorder (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast fibrosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast inflammation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast mass (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast necrosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Breast swelling (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cervical dysplasia (Reproductive system and breast disorders) | 2/2770 (2) | 0/2785 (0)
Endometrial disorder (Reproductive system and breast disorders) | 0/2770 (0) | 1/2785 (1)
Endometrial hypertrophy (Reproductive system and breast disorders) | 0/2770 (0) | 2/2785 (2)
Endometrial thickening (Reproductive system and breast disorders) | 1/2770 (1) | 1/2785 (1)
Endometriosis (Reproductive system and breast disorders) | 0/2770 (0) | 1/2785 (1)
Fibrocystic breast disease (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Metrorrhagia (Reproductive system and breast disorders) | 0/2770 (0) | 1/2785 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0/2770 (0) | 3/2785 (3)
Pelvic haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine polyp (Reproductive system and breast disorders) | 2/2770 (2) | 3/2785 (3)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 16 (16) | 3 (4)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 16 (17) | 3 (4)
Embolism (Vascular disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Lymphoedema (Vascular disorders) | 5 (5) | 3 (3)
Peripheral artery thrombosis (Vascular disorders) | 1 (1) | 1 (2)
Thrombophlebitis (Vascular disorders) | 2 (2) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 150 mg Abemaciclib + Endocrine Therapy (N=2791) | Endocrine Therapy (N=2800)
Anaemia (Blood and lymphatic system disorders) | 634 (862) | 88 (113)
Leukopenia (Blood and lymphatic system disorders) | 1026 (1706) | 171 (244)
Lymphopenia (Blood and lymphatic system disorders) | 372 (527) | 94 (118)
Neutropenia (Blood and lymphatic system disorders) | 1246 (2316) | 140 (214)
Thrombocytopenia (Blood and lymphatic system disorders) | 341 (528) | 39 (48)
Palpitations (Cardiac disorders) | 54 (62) | 20 (22)
Vertigo (Ear and labyrinth disorders) | 70 (93) | 47 (55)
Hypothyroidism (Endocrine disorders) | 28 (29) | 34 (34)
Dry eye (Eye disorders) | 71 (76) | 28 (31)
Lacrimation increased (Eye disorders) | 137 (158) | 10 (10)
Vision blurred (Eye disorders) | 46 (52) | 24 (25)
Abdominal distension (Gastrointestinal disorders) | 75 (90) | 27 (28)
Abdominal pain (Gastrointestinal disorders) | 945 (1974) | 226 (275)
Constipation (Gastrointestinal disorders) | 288 (377) | 142 (161)
Diarrhoea (Gastrointestinal disorders) | 2294 (11663) | 199 (288)
Dry mouth (Gastrointestinal disorders) | 94 (103) | 25 (27)
Dyspepsia (Gastrointestinal disorders) | 205 (264) | 61 (66)
Flatulence (Gastrointestinal disorders) | 84 (95) | 11 (12)
Gastritis (Gastrointestinal disorders) | 58 (65) | 31 (34)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 74 (76) | 45 (47)
Haemorrhoids (Gastrointestinal disorders) | 68 (82) | 28 (28)
Mouth ulceration (Gastrointestinal disorders) | 39 (48) | 3 (3)
Nausea (Gastrointestinal disorders) | 779 (1203) | 222 (274)
Stomatitis (Gastrointestinal disorders) | 154 (212) | 30 (39)
Toothache (Gastrointestinal disorders) | 49 (55) | 42 (50)
Vomiting (Gastrointestinal disorders) | 454 (744) | 117 (144)
Axillary pain (General disorders) | 28 (28) | 39 (41)
Chest pain (General disorders) | 35 (40) | 35 (36)
Chills (General disorders) | 49 (55) | 18 (18)
Fatigue (General disorders) | 1073 (1434) | 433 (522)
Influenza like illness (General disorders) | 141 (180) | 112 (152)
Malaise (General disorders) | 88 (109) | 29 (29)
Mucosal inflammation (General disorders) | 72 (90) | 21 (32)
Oedema peripheral (General disorders) | 169 (200) | 103 (119)
Pain (General disorders) | 60 (64) | 53 (58)
Peripheral swelling (General disorders) | 51 (58) | 53 (61)
Pyrexia (General disorders) | 227 (299) | 114 (130)
Hepatic steatosis (Hepatobiliary disorders) | 41 (42) | 35 (35)
Bronchitis (Infections and infestations) | 42 (50) | 40 (44)
Cellulitis (Infections and infestations) | 37 (43) | 28 (31)
Conjunctivitis (Infections and infestations) | 55 (63) | 30 (34)
Gastroenteritis (Infections and infestations) | 73 (84) | 32 (36)
Herpes zoster (Infections and infestations) | 34 (34) | 39 (39)
Influenza (Infections and infestations) | 110 (139) | 102 (135)
Nasopharyngitis (Infections and infestations) | 231 (324) | 186 (285)
Oral herpes (Infections and infestations) | 29 (34) | 8 (9)
Pharyngitis (Infections and infestations) | 26 (29) | 29 (33)
Pneumonia (Infections and infestations) | 45 (46) | 19 (19)
Sinusitis (Infections and infestations) | 69 (76) | 51 (67)
Skin infection (Infections and infestations) | 33 (36) | 23 (26)
Upper respiratory tract infection (Infections and infestations) | 280 (393) | 214 (323)
Urinary tract infection (Infections and infestations) | 278 (368) | 167 (235)
Vaginal infection (Infections and infestations) | 30/2770 (37) | 18/2785 (21)
Viral infection (Infections and infestations) | 28 (32) | 14 (15)
Vulvovaginal candidiasis (Infections and infestations) | 29/2770 (33) | 20/2785 (31)
Contusion (Injury, poisoning and procedural complications) | 42 (51) | 37 (38)
Fall (Injury, poisoning and procedural complications) | 52 (61) | 36 (43)
Procedural pain (Injury, poisoning and procedural complications) | 73 (78) | 53 (64)
Alanine aminotransferase increased (Investigations) | 265 (345) | 119 (149)
Aspartate aminotransferase increased (Investigations) | 257 (323) | 106 (122)
Blood alkaline phosphatase increased (Investigations) | 83 (98) | 47 (56)
Blood creatinine increased (Investigations) | 277 (396) | 17 (22)
Gamma-glutamyltransferase increased (Investigations) | 70 (80) | 24 (28)
Weight decreased (Investigations) | 79 (88) | 19 (20)
Weight increased (Investigations) | 29 (32) | 46 (47)
Decreased appetite (Metabolism and nutrition disorders) | 312 (352) | 54 (57)
Dehydration (Metabolism and nutrition disorders) | 33 (39) | 7 (7)
Hypercalcaemia (Metabolism and nutrition disorders) | 49 (58) | 32 (42)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 48 (53) | 61 (67)
Hyperglycaemia (Metabolism and nutrition disorders) | 37 (51) | 43 (53)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 67 (82) | 45 (63)
Hyperuricaemia (Metabolism and nutrition disorders) | 33 (44) | 13 (14)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 30 (39) | 12 (17)
Hypokalaemia (Metabolism and nutrition disorders) | 105 (126) | 22 (31)
Vitamin d deficiency (Metabolism and nutrition disorders) | 29 (33) | 33 (37)
Arthralgia (Musculoskeletal and connective tissue disorders) | 571 (705) | 876 (1117)
Arthritis (Musculoskeletal and connective tissue disorders) | 9 (10) | 29 (33)
Back pain (Musculoskeletal and connective tissue disorders) | 223 (277) | 271 (317)
Bone pain (Musculoskeletal and connective tissue disorders) | 62 (75) | 93 (102)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 24 (35) | 29 (40)
Joint stiffness (Musculoskeletal and connective tissue disorders) | 22 (25) | 56 (59)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 134 (180) | 100 (121)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 29 (31) | 16 (16)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 70 (77) | 72 (76)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 111 (120) | 154 (170)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 32 (34) | 33 (37)
Myalgia (Musculoskeletal and connective tissue disorders) | 167 (193) | 163 (185)
Neck pain (Musculoskeletal and connective tissue disorders) | 48 (49) | 59 (64)
Osteopenia (Musculoskeletal and connective tissue disorders) | 30 (30) | 32 (32)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 45 (45) | 71 (75)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 245 (292) | 274 (354)
Dizziness (Nervous system disorders) | 274 (333) | 158 (188)
Dysgeusia (Nervous system disorders) | 103 (121) | 8 (8)
Headache (Nervous system disorders) | 482 (809) | 359 (553)
Memory impairment (Nervous system disorders) | 29 (32) | 22 (22)
Neuropathy (Nervous system disorders) | 193 (221) | 203 (234)
Taste disorder (Nervous system disorders) | 36 (36) | 4 (4)
Anxiety (Psychiatric disorders) | 81 (84) | 113 (116)
Depression (Psychiatric disorders) | 134 (142) | 116 (120)
Insomnia (Psychiatric disorders) | 208 (251) | 218 (246)
Dysuria (Renal and urinary disorders) | 46 (53) | 25 (29)
Breast pain (Reproductive system and breast disorders) | 95 (104) | 120 (133)
Erectile dysfunction (Reproductive system and breast disorders) | 1/21 (1) | 0/15 (0)
Vaginal discharge (Reproductive system and breast disorders) | 26/2770 (27) | 39/2785 (42)
Vulvovaginal dryness (Reproductive system and breast disorders) | 78/2770 (80) | 117/2785 (127)
Cough (Respiratory, thoracic and mediastinal disorders) | 337 (407) | 193 (228)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 139 (154) | 77 (86)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 49 (52) | 8 (10)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 34 (37) | 29 (33)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 115 (142) | 76 (91)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 36 (36) | 10 (10)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 45 (53) | 25 (28)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 40 (41) | 40 (42)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 29 (31) | 15 (16)
Alopecia (Skin and subcutaneous tissue disorders) | 254 (266) | 53 (53)
Dermatitis (Skin and subcutaneous tissue disorders) | 28 (31) | 11 (13)
Dry skin (Skin and subcutaneous tissue disorders) | 102 (108) | 48 (51)
Eczema (Skin and subcutaneous tissue disorders) | 29 (32) | 28 (31)
Erythema (Skin and subcutaneous tissue disorders) | 38 (43) | 26 (28)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 29 (33) | 32 (34)
Nail disorder (Skin and subcutaneous tissue disorders) | 43 (45) | 4 (4)
Night sweats (Skin and subcutaneous tissue disorders) | 40 (43) | 28 (31)
Onychoclasis (Skin and subcutaneous tissue disorders) | 46 (54) | 7 (7)
Pruritus (Skin and subcutaneous tissue disorders) | 219 (298) | 110 (121)
Rash (Skin and subcutaneous tissue disorders) | 272 (332) | 106 (132)
Breast reconstruction (Surgical and medical procedures) | 28 (28) | 22 (25)
Hot flush (Vascular disorders) | 393 (432) | 587 (678)
Hypertension (Vascular disorders) | 101 (120) | 130 (158)
Hypotension (Vascular disorders) | 33 (33) | 14 (15)
Lymphoedema (Vascular disorders) | 282 (295) | 207 (225)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-09-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT03155997/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/97/NCT03155997/SAP_001.pdf